CLINICAL TRIAL: NCT07391124
Title: Pulp Temperature Elevation During Interproximal Reduction: An In Vivo Quantification of Temperature Changes Across Different Slenderization Methods
Brief Title: In Vivo Pulp Thermal Changes During Different Slenderization Techniques
Acronym: IPR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Alaina Tariq Mughal, Resident Orthodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 918/Trg
Record Dates: First submitted 2025-09-30; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Irreversible Pulpitis; Reversible Pulpitis; Thermal Injury; Pulp Hyperemia; Pulp Necrosis; Pulp Inflammation
Keywords: IPR; interproximal reduction; slenderization; thermal pulp damage; irreversible pulpitis; premolars; incisors
MeSH Terms: conditions — Dental Pulp Necrosis; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premolar Group (Experimental): Bilateral premolars planned for extraction as part of orthodontic treatment in a patient will undergo intervention using both the IPR methods to measure the changes in pup temperature. First baseline temperature wil be recorded intraorally then one side premolar (e.g; right) will undergo IPR using Air-rotor system and then the other side premolar (e.g; left) will undergo IPR using oscillating strip
  Interventions: Device: High-Speed Air-Driven Drill (Airotor and Bur); Device: Orthodontic IPR Kit (Oscillating System)
- Incisor Group (Experimental): Patients planned for lower single incisor extraction will be divided into two groups and undergo IPR using two different IPR techniques intraorally prior to extraction of the tooth.
  Interventions: Device: High-Speed Air-Driven Drill (Airotor and Bur); Device: Orthodontic IPR Kit (Oscillating System)

INTERVENTIONS:
Device: High-Speed Air-Driven Drill (Airotor and Bur) — This method involves high rotational speed (potentially over 300,000 RPM) and thus has the highest possibility of causing the greatest temperature elevation due to intense friction during interproximal reduction.
Device: Orthodontic IPR Kit (Oscillating System) — This technique operates at a much lower speed (around 5,000 RPM) and is expected to result in a moderate temperature increase, presenting a moderate possibility of thermal effect compared to the high-speed drill during interproximal reduction.

SUMMARY:
The goal of this study is to learn about the temperature rise inside the living part of a tooth (the pulp) during different ways of removing a small amount of enamel (the hard outer layer of the tooth), a procedure called Interproximal Enamel Reduction (IPR).

The goal of this study is to learn about the temperature rise inside the living part of a tooth (the pulp) during different ways of removing a small amount of enamel (the hard outer layer of the tooth), a procedure called Interproximal Enamel Reduction (IPR).

The main question it aims to answer is:

Which IPR technique causes the highest temperature rise in the live tooth pulp?

This study is important because, until now, no research has measured these temperature changes in the live pulp of teeth inside a person's mouth (in vivo) that includes both premolars and front teeth (incisors). The original studies only used premolars, and the results might be different for front teeth due to the difference in enamel thickness.

Researchers will use 20 premolar teeth and 20 incisors that will be scheduled for extraction as part of orthodontic treatment. The teeth will be divided into two groups based on the IPR method used:

Group 1: IPR using a high-speed air-driven drill (airotor) and bur. Group 2: IPR using an orthodontic IPR kit (an oscillating system).

Participants will:

Receive local anesthesia to numb the tooth. Have the baseline temperature of the pulp recorded using temperature sensor on either side of the teeth.

Have the temperature changes in the pulp recorded using temperature sensor while IPR is performed on the sides of the tooth.

Have the tooth extracted afterward (as part of original orthodontic plan)

The key findings may provide information of the IPR method that cause a temperature rise high enough to harm the pulp. A rise beyond 5.5∘C may cause pulp damage.

DETAILED DESCRIPTION:
Study Objectives The primary goal of this investigation is to evaluate the in vivo (inside the body) temperature rise within the dental pulp (the living tissue inside the tooth) when different techniques of Interproximal Enamel Reduction (IPR) are performed.

The core aims are:

1. To measure and compare the magnitude of pulp temperature increase across two common IPR methods.
2. To determine if any of the evaluated techniques have the potential to raise the pulp temperature above a critical threshold (5.5 degrees C), which is historically associated with irreversible pulp damage.
3. To identify which IPR technique carries the highest possibility of thermal injury.

Rationale and Significance Previous studies that looked at this issue were performed ex vivo (on extracted, non-living teeth). This study is crucial because it measures temperature changes in live, intact teeth under actual clinical conditions, providing a more reliable assessment of risk.

A key difference in this research, compared to other literature, is the inclusion of both incisors (front teeth) and premolars. Since the enamel thickness on incisors is generally less than on premolars, there is a possibility that the heat generated during IPR may transfer more readily to the pulp in the anterior teeth, potentially leading to a greater temperature rise and a higher risk of adverse thermal effects. This study aims to clarify this potential risk.

Study Design and Methods This is a randomized clinical trial, an in vivo study involving participants undergoing orthodontic treatment where tooth extraction is required.

Participant Population The study will involve participants for whom the extraction of specific teeth (premolars and incisors) has been clinically advised as part of their orthodontic treatment plan. These teeth will be used for the IPR procedures just before they are extracted.

Procedure Groups (Interventions)

The teeth will be randomly assigned to one of the following two IPR technique groups, with the potential for each to generate a different amount of frictional heat:

1. High-Speed Air-Driven Drill (Airotor and Bur): This method involves high rotational speed (potentially over 300,000 RPM) and thus has the highest possibility of causing the greatest temperature elevation due to intense friction.
2. Orthodontic IPR Kit (Oscillating System): This technique operates at a much lower speed (around 5,000 RPM) and is expected to result in a moderate temperature increase, presenting a moderate possibility of thermal effect compared to the high-speed drill.

Measurement Prior to the IPR procedure, local anesthesia will be administered. A sensitive thermocouple directly on the surface of tooth to meausre baseline temperature of the pulp.

The chosen IPR procedure will be performed. The temperature changes in the pulp will be monitored at two time points and recorded during the IPR process.

The data gathered will be used to compare the techniques and determine the relative possibility of thermal damage posed by each method, particularly within the incisors, which are uniquely included in this research.

ELIGIBILITY:
Inclusion Criteria:

* Participants 12 to 25 years of age.
* Participants undergoing orthodontic treatment requiring extraction of the teeth being studied (Incisors or Premolars).
* Selected tooth must be intact (no decay, large fillings, or fractures).
* Tooth must test vital (alive and healthy) prior to the procedure.
* Tooth must have healthy surrounding gum tissue.

Exclusion Criteria:

* Teeth that are non-vital (dead), have root canal treatment, or signs of irreversible pulpitis.
* Teeth with existing large or deep restorations (fillings) or crowns/veneers.
* Teeth that have undergone any previous IPR or stripping procedure.
* Teeth with significant developmental enamel defects (e.g., severe hypoplasia or fluorosis).
* Participants with severe systemic diseases (e.g., uncontrolled diabetes) affecting dental health.
* Participants taking medications that affect pulp sensation or vascular response (e.g., long-term anti-inflammatories).
* Participants who are pregnant or breastfeeding.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
The highest temperature reached inside the pulp chamber for each tooth during the IPR procedure | From enrollment to the date of planned extraction of the patient's teeth at 8 weeks so that all the measurements can be taken from T0 to T2 [T0 (prior to IPR procedure), TD (during IPR procedure with the techniques specified) T1 (immediately after IPR)]
  The highest temperature reached inside the pulp chamber for each tooth during the IPR procedure will be recorded using temperature sensor keeping it on the mid, mesial and distal facial surfaces of the tooth at different tie points; T0 (prior to IPR procedure), TD (during IPR procedure with the techniques specified) T1 (immediately after IPR), and T2 (after 5 mins post IPR)
Mean maximum temperature rise per IPR technique | from enrollment to the point of extraction of patient's teeth at 8 weeks
  Description: The calculated average of the maximum temperature rise for all teeth treated with a specific IPR technique.
  Analysis: This measure will be broken down by IPR technique and by tooth type (incisors vs. premolars).
  Conclusion: The method that consistently produces the lowest mean temperature rise across all groups is considered the most thermally conservative method.

SECONDARY OUTCOMES:
Residual Pulp Temperature Difference at 5 Minutes Post-IPR | From enrollment to the date of planned extraction of the patient's teeth at 8 weeks so that all the measurements can be taken from T0 to T2 [T0 (prior to IPR procedure), TD (during IPR procedure with the techniques specified) T1 (immediately after IPR)]
  The remaining temperature difference between the recorded pulp temperature at the 5-minute mark (T2) and the tooth's original baseline temperature (T0).
  This directly measures the thermal recovery efficiency of the tooth. A difference closer to 0∘ C will indicate faster and more complete recovery, suggesting the IPR technique/tooth type is better able to manage thermal stress.

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Tariq Mughal, BDS, FCPS (R), Principal Investigator — Armed Forces Institute of Dentistry, Pakistan
Locations (1):
- Armed Forces Intitute of Denistry (AFID), Combined Military Hospital (CMH), Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Conditions for Sharing:
  Request Process: Requests must be made formally to the Principal Investigator (or corresponding author) of the study.
  Purpose: Requests must include a detailed research proposal outlining the scientific rationale for using the data.
  Anonymization: All shared data will be fully anonymized to protect participant confidentiality and meet the requirements set forth by the institutional ethics review board.
  Timing: Data will be made available following the publication of the main study results.
  Data Use Agreement: Researchers accessing the data will be required to sign a formal data use agreement to ensure the data is used only for the approved purpose and is not shared further.

REFERENCES:
- See also: In vivo study measuring pulp ΔT during IPR with high-speed, oscillating, and manual methods on premolars. All methods were deemed thermally safe (ΔT<5.5 ∘C). This justifies extending the safety analysis to incisors. — https://rdcu.be/eIOLz